CLINICAL TRIAL: NCT02556437
Title: Randomized, Single-blind, Cross-over Study Investigating the Non-inferiority of Efficacy and Safety of HyQvia in Comparison With Conventional Subcutaneous Ig Therapy in Multifocal Motor Neuropathy
Brief Title: Efficacy and Safety of HyQvia (Immunoglobulin 10% With Recombinant Hyaluronidase) in Multifocal Motor Neuropathy (MMN)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johannes Jakobsen (Other)
Collaborators: Baxter Healthcare Corporation (Industry)
Responsible Party: Sponsor-Investigator, Johannes Jakobsen, Professor, DMSc, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: RH-2015-200
Record Dates: First submitted 2015-09-18; First posted 2015-09-22 (Estimated); Last update posted 2018-05-17 (Actual); Status verified 2018-05

CONDITIONS: Multifocal Motor Neuropathy
Keywords: Subcutaneous immunoglobulin; MMN
MeSH Terms: interventions — Immunoglobulins, Intravenous

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group A (Experimental): 24 weeks of treatment with conventional subcutaneous immunoglobulin (Subcuvia) followed by 24 weeks of treatment with HyQvia
  Interventions: Drug: HyQvia; Drug: Subcuvia
- Group B (Experimental): 24 weeks of treatment with HyQvia followed by 24 weeks of treatment with conventional subcutaneous immunoglobulin (Subcuvia)
  Interventions: Drug: HyQvia; Drug: Subcuvia

INTERVENTIONS:
Drug: HyQvia — Human immunoglobulin 10% with recombinant hyaluronidase for subcutaneous injection
  Other Names: Human immunoglobulin
Drug: Subcuvia — Human immunoglobulin 16% for subcutaneous injection
  Other Names: Human immunoglobulin

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of HyQvia (Immunoglobulin 10% with recombinant hyaluronidase) with conventional subcutaneous immunoglobulin treatment in patients with Multifocal Motor Neuropathy (MMN).

DETAILED DESCRIPTION:
Subcutaneous immunoglobulin (SCIG) therapy for MMN is equally efficacious to intravenous immunoglobulin (IGIV), may be self-induced and may induce fewer systemic adverse reactions. Limited SC infusion volumes and reduced bioavailability, however, necessitate multiple infusion sites, more frequent treatment, and dose adjustment to achieve pharmacokinetic equivalence. This is an issue in particular in MMN where relatively high and frequent doses are necessary to maintain long-term improvement of muscle strength. Recombinant human hyaluronidase (rHuPH20) increases subcutaneous tissue permeability and facilitates dispersion and absorption, enabling subcutaneous administration of higher (monthly) doses of Ig. If treatment with HyQvia is at least equally effective and safe as compared with conventional Ig treatment, HyQvia could become the preferred treatment option for patients with MMN as it may have attractive benefits for patients by its mode of administration.

ELIGIBILITY:
Inclusion Criteria:

* Age at onset 18 - 65 years.
* The presence of asymmetrical limb weakness at onset or motor involvement having a motor nerve distribution in at least two peripheral nerve distributions, predominant upper limb involvement, disabling weakness MRC grade 4 or less in at least one muscle.
* Decreased or absent tendon reflexes in affected limbs.
* Electrophysiological evidence of one site with definite motor conduction block or one site with probable conduction block according to previously defined criteria.
* Response to SCIG according to criteria that were described in previous studies
* On SCIG maintenance treatment for more than 3 months preceding the study.
* Patients have given written informed consent, prior to the study, with the understanding that consent may be withdrawn at any time without prejudice.

Exclusion Criteria:

* Bulbar signs or symptoms.
* Upper motor neuron signs (spasticity, hyperreflexia, extensor plantar response).
* Sensory symptoms and signs with sensory deficits on examination (except for vibration sense) and abnormal results of sensory nerve conduction studies
* Other neuropathies (e.g. diabetic, lead, porphyric or vasculitic neuropathy, chronic inflammatory demyelinating polyneuropathy, Lyme neuroborreliosis, post radiation neuropathy, hereditary neuropathy with liability to pressure palsies, Charcot-Marie-Tooth neuropathies, meningeal carcinomatosis).
* Treatment with other immunosuppressive drugs (cyclophosphamide, azathioprine, cyclosporin) in the 6 months preceding the study.
* Female patient who is pregnant or breast-feeding or of childbearing potential.
* Confirmation that the patient is not pregnant will be established by a negative b-HCG test within a 7-day period before inclusion in the study. Lack of childbearing potential is met by a) being post-menopausal, b) being surgically sterile, c) practising contraception with an oral contraceptive, intra-uterine device, diaphragm or condom with spermicide or d) being sexually inactive.
* Age < 18 years

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2016-06; Primary Completion 2018-05 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
Changes in isometric muscle strength | Evaluation at week 0, 12, 24, 36, 48
  Measurement of isometric muscle strength of four involved muscle groups

SECONDARY OUTCOMES:
Changes in disability score | Evaluation at week 0, 12, 24, 36, 48
  Disability are evaluated by the use of Guy´s Neurological Disability Scale
Changes in clinical evaluation of muscle strength | Evaluation at week 0, 12, 24, 36, 48
  Medical Research Council (MRC) sum score of 9 muscle groups bilateral (shoulder abduction, elbow flexion/extension, wrist flexion/extension, hip flexion, knee flexion/extension, ankle dorsal flexion)
Development of Headache and Nausea | During the entire study period
  Participants are asked to register severity of headache and nausea on a VAS scale from 0-100 mm on every day of infusion and the day after.
Development of hemolytic anemia | Evaluation at week 0, 12, 24, 36, 48
  Blood samples are drawn at every visit and are analyzed for hemoglobin and related parameters
Development of antibody against hyaluronidase | Evaluation at week 0, 12, 24, 36, 48
  Blood analyzed for specific antibodies against hyaluronidase
Patient satisfaction | Evaluation at week: 6, 12, 18, 24, 30, 36, 42, 48
  Patient are asked predefined question about satisfaction with the two treatment regimens and score them on a Visual Analogue Scale from 0-100 mm
Changes in grip strength | Evaluation at week 0, 12, 24, 36, 48
  Grip strength measured by Jamar® Hand dynamometer
Changes in hand/finger function | Evaluation at week 0, 12, 24, 36, 48
  9-hole peg test. Standardized test of hand/finger function.
Changes in gait performance | Evaluation at week 0, 12, 24, 36, 48
  40 meter walk test. Standardized test of walking performance.

CONTACTS AND LOCATIONS:
Overall Officials: Johannes Jakobsen, DMSc, Principal Investigator — Neuroscience Center, Rigshospitalet
Locations (2):
- Denmark (2):
  - Department of Neurology, Aarhus University Hospital, Aarhus C
  - Department of Neurology, Rigshospitalet, Copenhagen